CLINICAL TRIAL: NCT03697980
Title: Apogee, A HeartWare HVAD Destination Product Surveillance Registry (PSR) Platform
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: Apogee
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Results first posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- HVAD Left Ventricular Assist Device: Device: HeartWare Ventricular Assist Device
  Other Names:
  HVAD The HVAD is an implantable centrifugal rotary blood pump that is implanted in the pericardial space and is designed to provide up to 10 L/min of blood flow from the left ventricular to the aorta. The HVAD System is comprised of three major components: the HVAD (pump) with inflow and outflow conduits, a Controller (microprocessor unit that controls the operation of the HVAD), and power sources (AC and DC power adapters that provide power to the Controller and implanted HVAD).
  Interventions: Device: HeartWare Ventricular Assist Device

INTERVENTIONS:
Device: HeartWare Ventricular Assist Device — The HVAD is an implantable centrifugal rotary blood pump that is implanted in the pericardial space and is designed to provide up to 10 L/min of blood flow from the left ventricular to the aorta. The HVAD System is comprised of three major components: the HVAD (pump) with inflow and outflow conduits, a Controller (microprocessor unit that controls the operation of the HVAD), and power sources (AC and DC power adapters that provide power to the Controller and implanted HVAD).
  Other Names: HVAD

SUMMARY:
Medtronic is sponsoring the Apogee study to further enhance scientific understanding of the implant procedure, optimized blood pressure management, and anticoagulation/ antiplatelet therapy in patients receiving a Medtronic HeartWare™ Ventricular Assist Device (HVAD™) for destination therapy.

The Apogee study is conducted within Medtronic's Product Surveillance Platform.

DETAILED DESCRIPTION:
The Apogee study is a prospective, observational, post-market, on-label, multi-site study in Destination Therapy patients. Patients participating in the Medtronic Destination Therapy (DT) Post Approval Study (PAS) (NCT03681210) are eligible for participation in Apogee. Patients enrolled in Apogee will be followed under the Apogee study for one-year post-implant. After participation in Apogee ends, patients will remain enrolled in DT PAS and will continue to be followed as outlined in the DT PAS protocol. The total estimated study duration is 33 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects consented to participate in DT PAS are eligible for participation in Apogee.

Exclusion Criteria:

* There are no exclusion criteria unique to Apogee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in DT PAS (NCT03681210) are eligible for enrollment into Apogee and must be consented on the separate Apogee consent. It is expected that the Apogee cohort will be comprised of approximately 100 patients.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Saint Vincent Heart Clinic Arkansas, Little Rock, Arkansas
  - University of California San Diego, San Diego, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Stanford University Hospital, Stanford, California
  - University of Colorado, Aurora, Colorado
  - AdventHealth, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - Cardiac Surgery Clinical Research Center, Oak Lawn, Illinois
  - The University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Langone Medical Center, New York, New York
  - Columbia University, New York, New York
  - The Lindner Christ Hospital, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - University of Pittsburgh Medical Center UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Sciences Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwalth University Health System, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were considered enrolled upon signing informed consent. 12 enrolled participants weren't implanted due to death or screen failure prior to implant.
Groups:
- HVAD: HeartWare Ventricular Assist Device: The HVAD is an implantable centrifugal rotary blood pump that is implanted in the pericardial space and is designed to provide up to 10 L/min of blood flow from the left ventricular to the aorta. The HVAD System is comprised of three major components: the HVAD (pump) with inflow and outflow conduits, a Controller (microprocessor unit that controls the operation of the HVAD), and power sources (AC and DC power adapters that provide power to the Controller and implanted HVAD).
Period: Overall Study
Arm/Group | HVAD
Started | 124
Completed | 119
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: All implanted participants are included
Arm/Group | HVAD
Number analyzed (Participants) | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 103
  Unknown or Not Reported | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1
  Race: Asian | 3
  Race: Black or African American | 36
  Race: Native Hawaiian or Other Pacific Islander | 2
  Race: White | 73
  Race: Other | 9
Region of Enrollment [Number; unit: participants]
  United States | 124
Device Strategy at Time of Implant [Count of Participants; unit: Participants]
  Bridge to Transplant | 0
  Destination Therapy | 124

OUTCOME MEASURES:

1. Primary Outcome: Rate of Major Adverse Events
Description: Freedom from event is the probability (expressed as a percent of 100) the participant did not have a major adverse event during 12 months post implant via the Kaplan-Meier method. Participants that did not have a major adverse event were censored at the time of last follow-up in Apogee or their end of study at 12 months post implant, whichever occurred first.
  Major adverse events are defined to be occurrence of infection, bleeding, device malfunction, CT confirmed stroke, or death. Infection, bleeding, device malfunction and CT confirmed stroke were categorized via Intermacs Version 5.0.
  Events occurring during the implant procedure were excluded.
Time Frame: Implant to 12 months
Population: All implanted participants are included.
Measure: Number (95% Confidence Interval); unit: % probability of freedom from major AE
Arm/Group | HVAD
Number analyzed (Participants) | 124
% probability of freedom from major AE | 18.2 [11.8 to 25.8]

ADVERSE EVENTS:
Time Frame: The adverse events are summarized from the date of implant through 12 months while on the HVAD device. Only participants who are implanted with the device are included. All-cause mortality includes all participants who signed consent, regardless if they were implanted.
Description: The Intermacs adverse event definitions are geared towards participants who have a mechanical circulatory support device.
Arm/Group | HVAD
All-Cause Mortality (participants affected / at risk) | 27/136
Serious Adverse Events (participants affected / at risk) | 109/124
Other Adverse Events (participants affected / at risk) | 24/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HVAD (N=124)
Major Bleeding (Blood and lymphatic system disorders) | 54 (96)
Cardiac Arrhythmia (Cardiac disorders) | 40 (53)
Device Malfunction/Failure (Product Issues) | 12 (13)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Hepatic Dysfunction (Hepatobiliary disorders) | 6 (6)
Hypertension (Cardiac disorders) | 3 (4)
Infection (Infections and infestations) | 59 (95)
Myocardial Infarction (Cardiac disorders) | 0 (0)
Neurological Dysfunction (Nervous system disorders) | 30 (40)
Pericardial Fluid Collection (Cardiac disorders) | 3 (3)
Psychiatric Episode (Psychiatric disorders) | 11 (14)
Renal Dysfunction (Renal and urinary disorders) | 25 (28)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 20 (29)
Right Heart Failure (Cardiac disorders) | 33 (35)
Arterial Non-CNS Thromboembolism (Vascular disorders) | 2 (2)
Venous Thromboembolism (Vascular disorders) | 7 (7)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 0 (0)
Other Intermacs (General disorders) | 62 (155)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HVAD (N=124)
Infection (Infections and infestations) | 12 (13)
Other Intermacs (General disorders) | 16 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT03697980/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT03697980/SAP_001.pdf